CLINICAL TRIAL: NCT02256709
Title: Safety, Tolerability and Pharmacokinetics of BIBP 5371 CL Following Oral Administration to Healthy Male and Female Volunteers (Dose Range: 10 - 350 mg). A Double-blind (Within Treatment Groups), Randomised, Placebo-controlled, Single Rising Dose Study, Including Comparisons of 50 mg vs. 100 mg Tablet and Tablet vs. Drinking Solution, and Investigation of Food Effect
Brief Title: Safety, Tolerability and Pharmacokinetics of Oral BIBP 5371 CL in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1214.1
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets; Solutions

ARMS (8):
- single rising dose BIBP 5371 CL (Experimental)
  Interventions: Drug: BIBP 5371 CL tablet
- BIBP 5371 CL tablet high dose (Experimental): to be compared with same daily dose level from single rising dose arm
  Interventions: Drug: BIBP 5371 CL tablet high dose
- BIBP 5371 CL tablet low dose (Experimental): to be compared with same daily dose level from single rising dose arm
  Interventions: Drug: BIBP 5371 CL tablet low dose
- Placebo drinking solution (Placebo Comparator)
  Interventions: Drug: Placebo drinking solution
- BIBP 5371 CL drinking solution (Experimental)
  Interventions: Drug: BIBP 5371 CL solution
- BIBP 5371 CL tablet high dose with food (Experimental)
  Interventions: Other: High fat, high caloric breakfast; Drug: BIBP 5371 CL tablet high dose
- BIBP 5371 CL tablet low dose with food (Experimental)
  Interventions: Other: High fat, high caloric breakfast; Drug: BIBP 5371 CL tablet low dose
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: BIBP 5371 CL tablet — single rising daily doses
  Arms: single rising dose BIBP 5371 CL
Drug: BIBP 5371 CL solution
  Arms: BIBP 5371 CL drinking solution
Other: High fat, high caloric breakfast
  Arms: BIBP 5371 CL tablet high dose with food; BIBP 5371 CL tablet low dose with food
Drug: Placebo tablet
  Arms: Placebo tablet
Drug: BIBP 5371 CL tablet high dose
  Arms: BIBP 5371 CL tablet high dose; BIBP 5371 CL tablet high dose with food
Drug: Placebo drinking solution
  Arms: Placebo drinking solution
Drug: BIBP 5371 CL tablet low dose
  Arms: BIBP 5371 CL tablet low dose; BIBP 5371 CL tablet low dose with food

SUMMARY:
Safety, tolerability and pharmacokinetics (including comparisons of different formulations and investigation of food effect)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Age 21 - 50 years
* Body mass index (BMI) 18.5 - 29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, respiratory rate, body temperature and ECG) deviating from normal
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least 1 month or less than 10 half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial (within 1 week prior to administration or during the trial)
* Participation in another trial with an investigational drug (within 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 grams/day)
* Drug abuse
* Blood donation (≥ 100 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance

In addition, for female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraceptives, intrauterine device, sterilisation

Females, who are not surgically sterile will be asked to additionally use barrier contraception methods (e.g. condoms) prior to administration of study medication, during the study and at least 1 month after release from the study

* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2004-04; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with changes in vital signs | baseline, up to 8 days after drug administration
  blood pressure, pulse rate, respiratory rate, body temperature
Number of patients with changes in electrocardiogram (ECG) | baseline, up to 8 days after drug administration
Number of patients with changes in safety laboratory parameters | baseline, up to 8 days after drug administration
Number of patients with adverse events | baseline, up to 8 days after drug administration
Global tolerability assessment by the investigator on a verbal rating scale | up to 8 days after drug administration

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 32 hours after drug administration
tmax (time from dosing to maximum concentration) | up to 32 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 32 hours after drug administration
%AUC0-tz (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 32 hours after drug administration
λz (terminal rate constant in plasma) | up to 32 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 32 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 32 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 32 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 32 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 32 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 32 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 32 hours after drug administration